CLINICAL TRIAL: NCT06052722
Title: The Relationship of Premenstrual Syndrome and Primary Dysmenorrhea With Severity of Temporomandibular Disorders
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Tokat Gaziosmanpasa University (Other)
Responsible Party: Principal Investigator, Halime Arikan, Assistant Professor, Tokat Gaziosmanpasa University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: 13.21
Record Dates: First submitted 2023-09-13; First posted 2023-09-25 (Actual); Last update posted 2023-09-25 (Actual); Status verified 2023-09

CONDITIONS: Primary Dysmenorrhea; Premenstrual Syndrome; Temporomandibular Disorder
Keywords: Primary Dysmenorrhea; Premenstrual Syndrome; Temporomandibular Disorder; Correlation; Relationship
MeSH Terms: conditions — Premenstrual Syndrome; Temporomandibular Joint Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Individuals with premenstrual syndrome (Other): Level of relationship between premenstrual syndrome and temporomandibular disorders
  Interventions: Other: Correlation assessment
- Individuals with primary dysmenorrhea (Other): Level of relationship between primary dysmenorrhea and temporomandibular disorders
  Interventions: Other: Correlation assessment

INTERVENTIONS:
Other: Correlation assessment — The relationship between the Premenstrual Syndrome Impact Scale and the Fonseca Anamnestic Index will be examined for individuals with premenstrual syndrome. The relationship between Working Ability, Location, Intensity, Days of Pain, Dysmenorrhea Score and Fonseca Anamnestic Index will be examined for individuals with primary dysmenorrhea.

SUMMARY:
Premenstrual pain, menstrual pain, other pains, and somatic symptoms may occur together. Therefore, this study aims to examine the severity of temporomandibular disorders in individuals complaining of premenstrual syndrome or dysmenorrhea and its relationship.

DETAILED DESCRIPTION:
The sample of the study will consist of at least 60 adult female individuals over the age of 18 with premenstrual syndrome or primary dysmenorrhea residing in Tokat. Premenstrual Dysphoria Disorder DSM-5 Diagnostic Criteria will be used to determine the presence of premenstrual syndrome. In cases of classic primary dysmenorrhea, a pelvic examination is not necessary to begin treatment. There is no specific test to identify primary dysmenorrhea, but individuals with the classic presentation are candidates for empiric therapy. These individuals were identified according to the following characteristics: 1) Menstrual pain that begins within a few months or within 2 years after menarche, 2) Pain that begins just before or at the beginning of menstruation, 3) Pain that can radiate to the lower abdomen and back, inner thighs, or both, 4) ) Pain that rarely lasts more than 72 hours, 5) Episodic and cramp-like pain, 6) Similar pain from one menstrual cycle to the next, and 7) Additional symptoms such as nausea and vomiting, fatigue, headache, dizziness and sleep disturbances. To exclude secondary dysmenorrhea: 1) Dysmenorrhea occurring during the first one or two cycles after menarche, 2) Dysmenorrhea starting after the age of 25, 3) Late onset of dysmenorrhea after a history of no pain with menstruation, 4) Infertility (endometriosis, pelvic inflammatory disease). ), heavy menstrual flow, or irregular cycles (adenomyosis, fibroids, polyps), individuals with dyspareunia will be recorded as secondary dysmenorrhea and excluded from the study. In line with these criteria, an inquiry will be made and appropriate individuals will be included in the study. In this study, power analysis was performed with the G*Power program to determine the sample size. Taking the type one error as (α)=0.05, the power of the study as (β)=0.95, the acceptable correlation rate as (r)=0.70, and the negligible correlation rate as (r)=0.30, the sample required to determine the relationship between premenstrual syndrome and temporomandibular disorders severity was determined. The size was calculated as 30 participants. Likewise, 30 participants will be required to determine the relationship between dysmenorrhea and temporomandibular disorders severity. Therefore, the number of individuals required to participate in this study was calculated as 60. After individuals' sociodemographic information is questioned, data will be collected with other outcome measurements. Individuals will be invited verbally to the study and a face-to-face survey will be administered to those who volunteer.

ELIGIBILITY:
Inclusion Criteria:

* To be volunteer

Exclusion Criteria:

* Having any gynecological or obstetric diagnosis other than premenstrual syndrome or primary dysmenorrhea
* Being pregnant
* Having any neurological, psychiatric or cognitive disorder.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-10-01 (Estimated); Primary Completion 2023-12-01 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Premenstrual Syndrome Impact Scale | up to 3 months
  The Premenstrual Syndrome Impact Scale consists of 18 items. It assesses psychological stress and functional interaction in daily life and is designed for premenstrual symptoms. It considers the complex and multifaceted nature of the disorder, thus facilitating the diagnosis process by assessing the necessary impact and enabling the planning and evaluation of treatment. It has a 4-point Likert-type answering system. Increasing the score means that the exposure increases. The questionnaire is valid and reliable in the Turkish population.
Working Ability, Location, Intensity, Days of Pain, Dysmenorrhea Score | up to 3 months
  Working Ability, Location, Intensity, Days of Pain, Dysmenorrhea Score consists of 4 items. It was designed as a scale-type questionnaire integrating dysmenorrhea features: 1) Number of anatomical pain locations (no part of the body, lower abdomen, lumbar area, lower extremities, groin area), 2) Wong-Baker pain rating (doesn't hurt, hurts a little, hurts a little more, hurts a lot, hurts more, hurts a lot, hurts a lot), 3) Number of painful days during the menstrual period (0, 1-2, 3-4, ≥5) and 4) Frequency of pain that prevents performing activities (never, almost never, almost always, always). Each item has a score between 0 and 3. The total score varies between 0 and 12 points. An increasing score indicates a greater degree of dysmenorrhea. The scale is valid and reliable in Turkish population.
Fonseca Anamnestic Index | up to 3 months
  The presence and severity of temporomandibular disorders in individuals will be questioned with the Fonseca Anamnestic Index. The Fonseca Anamnestic Index consists of 10 questions. The participant is asked to answer each question as 'Yes' (10 points), 'No' (0 points), and 'Sometimes' (5 points). The questionnaire score is scored for all questions, and temporomandibular disorder severity is classified according to the total score: no temporomandibular disorder (0-15 points), mild temporomandibular disorder (20-40 points), moderate temporomandibular disorder (45-65 points), severe temporomandibular disorder (70-100). Turkish version validity and reliability study was conducted.

CONTACTS AND LOCATIONS:
Locations (1):
- Tokat Gaziosmanpasa University, Tokat Province, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided